CLINICAL TRIAL: NCT04226755
Title: Liberal Use of Sodium in Ambulatory Heart Failure
Acronym: LUSA-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, Principal investigator, Ziekenhuis Oost-Limburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZOLCAR19001
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: Sodium; Salt; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure (Experimental): After a run-in phase of 2 weeks, patients will add 3 g of sodium chloride to every meal, using a NaCl tablet of 1 g. They will continue the sodium tablet for 4 weeks with a study visit every 2 weeks. A skin biopsy will be performed before the start of the augmented salt intake and after 4 weeks.
  Interventions: Dietary Supplement: Sodium chloride
- Healthy volunteer (Active Comparator): After a run-in phase of 2 weeks, volunteers will add 3 g of sodium chloride to every meal, using a NaCl tablet of 1 g. They will continue the sodium tablet for 4 weeks with a study visit every 2 weeks.A skin biopsy will be performed before the start of the augmented salt intake and after 4 weeks.
  Interventions: Dietary Supplement: Sodium chloride

INTERVENTIONS:
Dietary Supplement: Sodium chloride — 1 gram tid (with every meal)

SUMMARY:
This study investigates the effects of an increased sodium intake in heart failure patients with reduced ejection fraction and age-matched volunteers without heart failure.

DETAILED DESCRIPTION:
At the start of the study, baseline investigations are performed including assessment of vital signs (blood pressure, heart rate, pulse oxygen saturation), weight, Everest congestion score (consisting of grading of dyspnea, orthopnea, jugular venous distention, rales, edema and fatigue), echocardiography, 24h urine collection, bio-impedance measurements and blood sample analysis with plasma renin and aldosterone Subsequently, a run-in phase of 2 weeks, without intervention, will start. After this run-in period, participants will be reassessed with the same baseline investigations. In addition, a skin biopsy will be performed as well as a blood volume measurement.

In the next phase of the study, salt intake will be increased with 3 grams daily. The salt will be packed in capsules containing 1 g of sodium chloride (NaCl). Patients will be asked to take one capsule with their breakfast, lunch and dinner. Every 2 weeks a follow-up visit is planned.

After 4 weeks of increased salt intake, a new skin biopsy will be taken and a blood volume measurement will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Heart failure patients:

   * Left ventricular ejection fraction ≤40% on echocardiogram obtained at inclusion
   * Stable dose of guideline-recommended disease modifying drugs for at least 3 months.
   * Maximum daily loop diuretic dose of 40 mg furosemide equivalents with a stable dose for the last month
2. Healthy volunteers:

   * Age > 60 y
   * Normal ejection fraction (>50%) without heart failure
   * No neurohormonal blockers for hypertension
   * Normal NT-proBNP

Exclusion Criteria:

* Heart failure hospitalization for congestion or myocardial infarction in past 3 months
* Permanent atrial fibrillation
* New York Heart Association (NYHA) class III-IV
* Estimated glomerular filtration rate (eGFR) < 30 mL/min
* Signs of congestion
* Severe right ventricular dysfunction
* Severe valvular disease
* Cardiothoracic anatomy not allowing satisfactory and reproducible recordings of echocardiogram
* Inability to fully comprehend and/or perform study procedures in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in skin glycosaminoglycan (GAG) content | 4 weeks
Changes in skin sodium content | 4 weeks

SECONDARY OUTCOMES:
Changes in blood volume assessed by radiolabeled red blood cell technique | 4 weeks
Changes in extracellular, intravascular volume and total body fluid volume (assessed with bioimpedance) | 6 weeks
Changes in renal sodium handling | 6 weeks
Changes in cardiac geometry assessed by echo | 6 weeks
Changes in renal venous flow pattern | 6 weeks

OTHER OUTCOMES:
Changes in Everest congestion score | 6 weeks
  The Everest score assesses congestion, based on a point scale with a range from 0 (no congestion) to 18 (worst congestion)
Changes in weight | 6 weeks
Changes in blood pressure | 6 weeks
Changes in thirst visual analogue scale (VAS) | 6 weeks
  The scale ranges from 0 -100 with 0 indicating no thirst and 100 the worst thirst.
Changes in aldosterone | 6 weeks
Changes in renin | 6 weeks
Changes in N-terminal (NT)-pro hormone BNP (NT-proBNP) | 6 weeks
  NT-proBNP will be measured using Roche diagnostics assay (Mannhein, Germany) and expresed as picogram per liter
Occurrence of congestion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Dauw, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium